CLINICAL TRIAL: NCT03287817
Title: A Single Arm, Open-label, Multi-centre, Phase I/II Study Evaluating the Safety and Clinical Activity of AUTO3, a CAR T Cell Treatment Targeting CD19 and CD22 With Anti Programmed Cell Death Protein 1 (PD1) Antibody in Patients With Relapsed or Refractory Diffuse Large B Cell Lymphoma
Brief Title: Cluster of Differentiation Antigen 19/22(CD19/22) CAR T Cells (AUTO3) for the Treatment of Diffuse Large B Cell Lymphoma
Acronym: ALEXANDER
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: After reviewing the data and taking into consideration the available treatment landscape in r/r DLBCL, Autolus didn't progress into the Phase II part of the study and submitted a Notification of End of Trial (MHRA reference 46113/0003/001-0016).
Sponsor: Autolus Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AUTO3-DB1; 2016-004682-11 (EudraCT Number)
Record Dates: First submitted 2017-09-11; First posted 2017-09-19 (Actual); Results first posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-06

CONDITIONS: Relapsed/Refractory Diffuse Large B-Cell Lymphoma (DLBCL)
Keywords: Diffuse Large B Cell Lymphoma; Relapsed Diffuse Large B Cell Lymphoma; Refractory Diffuse Large B Cell Lymphoma; AUTO3; PD-1; Anti PD-1 antibody
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Intervention Model Description: A dose escalation and expansion phase (Phase I) followed by Phase II
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AUTO3 (Experimental): Patient with relapsed or refractory DLBCL
  Interventions: Biological: AUTO3

INTERVENTIONS:
Biological: AUTO3 — Following preconditioning with chemotherapy (cyclophosphamide and fludarabine) patients will be treated with doses from 50 x 10⁶ to 900 x 10⁶ CD19/ CD22 Chimeric Antigen Receptor (CAR) positive T cells with limited duration of anti-PD1 antibody (pembrolizumab).

SUMMARY:
The purpose of this study is to test the safety and efficacy of AUTO3, a CAR T cell treatment targeting CD19 and CD22 with consolidation or pre-conditioning with anti-PD1 antibody in patients with DLBCL

DETAILED DESCRIPTION:
The study will consist of 2 phases, a Phase I or dose escalation and expansion phase, and a Phase II. Patients with relapsed or refractory DLBCL will be enrolled in both phases of the study. Eligible patients will undergo leukapheresis in order to harvest T cells, which is the starting material for the manufacture of the autologous CAR T product AUTO3, a CD19 and CD22 dual targeting CAR T cell product. Following pre-conditioning by a chemotherapeutic regimen, the patient will receive AUTO 3 intravenously as a single dose and in addition a limited duration of treatment with an anti-PD1 antibody (either as part of the pre-conditioning regimen or consolidation). Patients will then enter a 36-month follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged ≥18 years.
2. Willing and able to give written, informed consent.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status 0 to 1.
4. Histologically confirmed DLBCL and large B cell lymphoma subsets, including:

   Phase I and Phase II Cohort 1:
   1. DLBCL, not otherwise specified (NOS), per World Health Organisation classification and DLBCL with MYC oncogene (MYC) and B cell lymphoma 2 (BCL2) gene and/or B cell lymphoma 6 (BCL6) gene rearrangements (double/triple hit).
   2. Transformed DLBCL from follicular lymphoma (FL).
   3. High-grade B cell lymphoma with MYC expression (excluding Burkitt's lymphoma) Phase I and Phase II Cohort 2.
   4. Transformed DLBCL from other indolent lymphomas (excluding Richter's transformation).
   5. Primary mediastinal large B cell lymphoma.
5. Chemotherapy-refractory disease, defined as one or more of the following:

   1. Stable disease (≤12 months) or progressive disease as best response to most recent chemotherapy containing regimen. Refractory disease after frontline chemo-immunotherapy is allowed.
   2. Disease progression or recurrence in ≤12 months of prior autologous haematopoietic stem cell transplantation (ASCT).

   OR
6. Relapse after ≥two lines of therapy or after ASCT. At a minimum:

   1. Patients must have received rituximab or another anti-cluster of differentiation antigen 20 (CD20) monoclonal antibody (unless Investigator determines that tumour is CD20-negative) and an anthracycline-containing chemotherapy regimen.
   2. Patients must have either failed ASCT, or be ineligible for or not consenting to ASCT.
   3. Patients with transformed DLBCL must have received at least one line of therapy after transformation to DLBCL.
7. Positron emission tomography-positive disease per Lugano classification.
8. For females of childbearing potential, a negative serum or urine pregnancy test must be documented at screening, prior to pre-conditioning and confirmed before receiving the first dose of study treatment.

   For females who are not postmenopausal or surgically sterile, highly effective methods of contraception must be used during the treatment period and for at least 12 months after the last dose of study treatment.
9. For males, it must be agreed that that two acceptable methods of contraception are used.
10. Adequate renal, hepatic, pulmonary, and cardiac function defined as:

    1. Creatinine clearance ≥40 cc/min.
    2. Serum alanine aminotransferase / aspartate aminotransferase ≤2.5 x upper limit of normal (ULN).
    3. Total bilirubin ≤1.5 x ULN, except in subjects with Gilbert's syndrome.
    4. Left ventricular ejection fraction (LVEF) ≥50% (by echocardiogram [ECHO] or Multiple gated acquisition scan [MUGA]) unless the institutional lower limit of normal is lower.
    5. Baseline oxygen saturation >92% on room air and ≤Grade 1 dyspnoea.
11. Patient has adequate bone marrow (BM) function without requiring ongoing blood product or granulocyte-colony stimulating factor support and meets the following criteria:

    1. Absolute neutrophil count ≥1.0 × 10^9/L.
    2. Absolute lymphocyte count ≥0.3 × 10^9/L (at enrolment and prior to leukapheresis).
    3. Haemoglobin ≥80 g/L.
    4. Platelets ≥75 × 10^9/L
12. No contra-indications for leukapheresis.

Exclusion Criteria:

1. Prior allogeneic haematopoietic stem cell transplant.
2. Females who are pregnant or lactating.
3. History or presence of clinically relevant CNS pathology such as epilepsy, paresis, aphasia, stroke within prior 3 months, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, uncontrolled mental illness, or psychosis.
4. Patients with active CNS involvement by malignancy. Patients with history of central nervous system (CNS) involvement with malignancy may be eligible if CNS disease has been effectively treated and provided treatment was at least 4 weeks prior to enrolment (at least 8 weeks prior to AUTO3 infusion).
5. Clinically significant, uncontrolled heart disease or a recent (within 12 months) cardiac event.

   1. Uncontrolled cardiac arrhythmia (patients with rate-controlled atrial fibrillation are not excluded).
   2. Evidence of pericardial effusion
6. Patients with a history (within 3 months) or evidence of deep vein thrombosis or pulmonary embolism requiring ongoing therapeutic anticoagulation at the time of pre-conditioning.
7. Patients with active gastrointestinal bleeding.
8. Patients with any major surgical intervention in the last 3 months.
9. Active bacterial, viral or fungal infection requiring systemic treatment. Active or latent hepatitis B infection or hepatitis C infection. Testing positive for human immunodeficiency virus, human T cell lymphotropic virus (HTLV1 and 2) or syphilis.
10. History of autoimmune disease resulting in end organ injury or requiring systemic immunosuppression/systemic disease modifying agents within the last 24 months.
11. Patients with a known history or prior diagnosis of optic neuritis or other immunologic or inflammatory disease affecting the CNS.
12. Evidence of active pneumonitis on chest computed tomography (CT) scan at screening or history of drug-induced pneumonitis, idiopathic pulmonary fibrosis, organising pneumonia, or idiopathic pneumonitis.
13. History of other malignant neoplasms unless disease free for at least 24 months (carcinoma in situ, non-melanoma skin cancer, breast or prostate cancer on hormonal therapy allowed).
14. Prior treatment with PD1, programmed cell death ligand 1 (PD-L1), or cytotoxic T lymphocyte-associated protein-4-targeted therapy, or tumour necrosis factor (TNF) receptor superfamily agonists within 6 weeks prior to AUTO3 infusion.
15. Prior treatment with investigational or approved gene therapy or cell therapy products until a dose level has treated at least three patients and has been declared safe.
16. Prior CD19 or CD22 targeted therapy.
17. The following medications are excluded:

    1. Steroids: Therapeutic doses of corticosteroids within 7 days of leukapheresis or 72 hours prior to AUTO3 administration. However, physiological replacement, topical, and inhaled steroids are permitted.
    2. Immunosuppression: Immunosuppressive medication must be stopped ≥2 weeks prior to leukapheresis or AUTO3 infusion.
    3. Cytotoxic chemotherapies within 2 weeks of AUTO3 infusion and 1 week prior to leukapheresis (2 weeks for lymphodepleting chemotherapy).
    4. Antibody therapy use including anti-CD20 therapy within 2 weeks prior to AUTO3 infusion, or 5 half-lives of the respective antibody, whichever is shorter.
    5. Granulocyte-colony stimulating factor less than 10 days prior to leukapheresis.
    6. Live vaccine ≤4 weeks prior to enrolment.
    7. Prophylactic intrathecal therapy: Methotrexate within 4 weeks and other intrathecal chemotherapy (e.g. Ara-C) within 2 weeks prior to starting pre-conditioning chemotherapy.
18. Prior limited radiation therapy within 4 weeks of AUTO3 infusion or within 24 weeks for definitive radiation to chest.
19. Research participants receiving any other investigational agents, or concurrent biological, chemotherapy, or radiation therapy.
20. Known allergy to albumin, dimethyl sulphoxide (DMSO), cyclophosphamide or fludarabine, pembrolizumab or tocilizumab.
21. Any contraindications to receive anti-PD1 antibody pembrolizumab will be excluded from cohorts requiring administration of pembrolizumab.
22. Patients, who in the opinion of the Investigator, may not be able to understand or comply with the safety monitoring requirements of the study.
23. Any other condition that in the Investigator's opinion would make the patient unsuitable for the clinical trial.

    Phase I outpatient cohort:
24. Subjects who do not have caregiver support (in line with institutional outpatient transplant guidelines) for outpatient/ambulatory care setting.
25. Subjects who are staying greater than 60 minutes (or whatever is permissible per institutional outpatient transplant guidelines) from the clinical trial site at the time of treatment.

For AUTO3 Infusion: Patients meeting any of the following exclusion criteria must not be treated with AUTO3 or have treatment delayed until they no longer meet these criteria:

1. Severe intercurrent infection.
2. Requirement for supplementary oxygen or active pulmonary infiltrates.
3. Clinical deterioration of organ function (renal and hepatic) exceeding the criteria set at study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2023-10-19 (Actual); Study Completion 2023-10-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (7):
  - City of Hope Hospital, Duarte, California
  - Colorado Blood Cancer Institute at Presbyterian/St. Luke's Medical Center/Sarah Cannon Research Institute, Denver, Colorado
  - Sylvester Comprehensive Cancer Center / University of Miami, Miami, Florida
  - Siteman Cancer Center / Washington University School of Medicine, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - TriStar Centennial Medical Center /Sarah Cannon Research Institute, Nashville, Tennessee
  - St David's South Austin Medical Center /Sarah Cannon Research Institute, Austin, Texas
- United Kingdom (4):
  - The Beatson West of Scotland Cancer Centre / Queen Elizabeth University Hospital, Glasgow
  - University College London Hospitals NHS Foundation Trust, London
  - Manchester University NHS Foundation Trust, Manchester
  - Freeman Hospital, The Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne

REFERENCES:
- [Result] Roddie C, Lekakis LJ, Marzolini MAV, Ramakrishnan A, Zhang Y, Hu Y, Peddareddigari VGR, Khokhar N, Chen R, Basilico S, Raymond M, Vargas FA, Duffy K, Brugger W, O'Reilly MA, Wood L, Linch DC, Peggs KS, Bachier C, Budde EL, Lee Batlevi C, Bartlett N, Irvine D, Tholouli E, Osborne W, Ardeshna KM, Pule MA. Dual targeting of CD19 and CD22 with bicistronic CAR-T cells in patients with relapsed/refractory large B-cell lymphoma. Blood. 2023 May 18;141(20):2470-2482. doi: 10.1182/blood.2022018598. PMID 36821767
- [Derived] Ernst M, Oeser A, Besiroglu B, Caro-Valenzuela J, Abd El Aziz M, Monsef I, Borchmann P, Estcourt LJ, Skoetz N, Goldkuhle M. Chimeric antigen receptor (CAR) T-cell therapy for people with relapsed or refractory diffuse large B-cell lymphoma. Cochrane Database Syst Rev. 2021 Sep 13;9(9):CD013365. doi: 10.1002/14651858.CD013365.pub2. PMID 34515338

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 73 adult patients with r/r DLBCL were screened and 62 patients were enrolled. For these 62 patients AUTO3 was manufactured using leukapheresed autologous peripheral blood mononuclear cells, modified with a bicistronic transgene. Ten patients did not receive AUTO3 infusion, in 6 patients this was due to death, in 3 patients due to progressive disease (without death), and in 1 patient due to failed eligibility.
Groups:
- 50 x 10^6 Cluster of Differentiation Antigen 19/22 (CD19/CD22) CAR+ T Cells: Patients in this cohort received actual doses of 50 to 150 x 10^6 CD19/CD22 CAR+ T cells
- 50 x 10^6 CD19/CD22 CAR+ T Cells + Pembrolizumab at Day 14: Patients in this cohort received actual dose of 50 x 10^6 CD19/CD22 CAR+ T cells
- 150 to 450 x 10^6 CD19/CD22 CAR+ T Cells + Pembrolizumab at Day 14: Patients in this cohort received actual doses of 150 to 495 x 10^6 CD19/CD22 CAR+ T cells
- 150 to 450 x 10^6 CD19/CD22 CAR+ T Cells + Pembrolizumab at Day -1 in an Inpatient Setting: Patients in this cohort received actual doses of 125 to 450 x 10^6 CD19/CD22 CAR+ T cells + pembrolizumab at Day -1 in an inpatient setting
- 150 to 450 x 10^6 CD19/CD22 CAR+ T Cells + Pembrolizumab at Day -1 in an Outpatient Setting: Patients in this cohort received actual doses of 129 to 450 x 10^6 CD19/CD22 CAR+ T cells + pembrolizumab at Day -1 in an outpatient setting
Period: Overall Study
Arm/Group | 50 x 10^6 Cluster of Differentiation Antigen 19/22 (CD19/CD22) CAR+ T Cells | 50 x 10^6 CD19/CD22 CAR+ T Cells + Pembrolizumab at Day 14 | 150 to 450 x 10^6 CD19/CD22 CAR+ T Cells + Pembrolizumab at Day 14 | 150 to 450 x 10^6 CD19/CD22 CAR+ T Cells + Pembrolizumab at Day -1 in an Inpatient Setting | 150 to 450 x 10^6 CD19/CD22 CAR+ T Cells + Pembrolizumab at Day -1 in an Outpatient Setting
Started | 4 | 3 | 8 | 17 | 20
Completed | 0 | 1 | 3 | 3 | 4
Not Completed | 4 | 2 | 5 | 14 | 16
Not completed — Progressive disease | 4 | 2 | 3 | 10 | 8
Not completed — Death | 0 | 0 | 2 | 3 | 4
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Population: Sixty-two patients were enrolled. Ten patients did not receive AUTO3 infusion, in 6 patients this was due to death, in 3 patients due to progressive disease (without death), and in 1 patient due to failed eligibility, leaving 52 participants.
Groups:
- 50 x 10^6 Cluster of Differentiation (CD) 19/CD22 CAR-positive T Cells: Patients in this cohort received actual doses of 50 to 150 x 10^6 CD19/CD22 CAR-positive T cells
- 50 x 10^6 CD19/CD22 CAR-positive T Cells + Pembrolizumab at Day 14: All patients in this cohort received actual dose of 50 x 10^6 CD19/CD22 CAR-positive T cells + pembrolizumab at Day 14
- 150 to 450 x 10^6 CD19/CD22 CAR-positive T Cells + Pembrolizumab at Day 14: Patients in this cohort received actual doses of 150 to 495 x 10^6 CD19/CD22 CAR-positive T cells + pembrolizumab at Day 14
- 150 to 450 x 10^6 CD19/CD22 CAR-positive T Cells + Pembrolizumab at Day -1 in an Inpatient Setting: Patients in this cohort received actual doses of 125 to 450 x 10^6 CD19/CD22 CAR-positive T cells + pembrolizumab at Day -1 in an inpatient setting
- 150 to 450 x 10^6 CD19/CD22 CAR-positive T Cells + Pembrolizumab at Day -1 in an Outpatient Setting: Patients in this cohort received actual doses of 129 to 450 x 10^6 CD19/CD22 CAR-positive T cells + pembrolizumab at Day -1 in an outpatient setting
- Total: Total of all reporting groups
Arm/Group | 50 x 10^6 Cluster of Differentiation (CD) 19/CD22 CAR-positive T Cells | 50 x 10^6 CD19/CD22 CAR-positive T Cells + Pembrolizumab at Day 14 | 150 to 450 x 10^6 CD19/CD22 CAR-positive T Cells + Pembrolizumab at Day 14 | 150 to 450 x 10^6 CD19/CD22 CAR-positive T Cells + Pembrolizumab at Day -1 in an Inpatient Setting | 150 to 450 x 10^6 CD19/CD22 CAR-positive T Cells + Pembrolizumab at Day -1 in an Outpatient Setting | Total
Number analyzed (Participants) | 4 | 3 | 8 | 17 | 20 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 7 | 7 | 16 | 37
  >=65 years | 0 | 0 | 1 | 10 | 4 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 7 | 7 | 16 | 35
  Male | 2 | 0 | 1 | 10 | 4 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 5 | 6
  Not Hispanic or Latino | 4 | 3 | 8 | 16 | 9 | 40
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 6 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 3 | 4
  White | 4 | 3 | 8 | 15 | 14 | 44
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 3 | 3
Eastern Cooperative Oncology Group (ECOG) score [Count of Participants; unit: Participants] — 0 = Fully active, able to carry on all pre-disease performance without restriction; 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  Participants
    ECOG = 0 | 1 | 1 | 7 | 9 | 8 | 26
    ECOG = 1 | 3 | 2 | 1 | 8 | 12 | 26
Disease stage [Count of Participants; unit: Participants] — Positron emission tomography (PET), CT and MRI were used to determine disease stage at screening.
  Stage I - In 1 lymph region only or single extranodal site Stage II - In ≥ 2 lymph regions on the same side of the diaphragm, and may include limited contiguous extranodal involvement Stage III - In the lymph nodes, spleen, or both and on both sides of the diaphragm Stage IV - Extranodal involvement (eg, bone marrow, lungs, liver)
  Participants
    Stage II | 0 | 0 | 1 | 2 | 3 | 6
    Stage III | 0 | 2 | 2 | 3 | 4 | 11
    Stage IV | 4 | 1 | 5 | 12 | 13 | 35
Relapsed/Refractory disease [Count of Participants; unit: Participants]
  Relapsed | 0 | 0 | 1 | 4 | 11 | 16
  Refractory | 0 | 1 | 2 | 6 | 3 | 12
  Relapsed and Refractory | 4 | 2 | 5 | 7 | 6 | 24
Extranodal disease present [Count of Participants; unit: Participants]
  No | 2 | 2 | 3 | 6 | 7 | 20
  Yes | 2 | 1 | 5 | 11 | 13 | 32
Current lymphoma subtype [Count of Participants; unit: Participants]
  Non-Germinal center B cell type | 1 | 0 | 1 | 2 | 3 | 7
  Germinal center B cell type | 0 | 0 | 4 | 11 | 9 | 24
  Activated B cell type | 2 | 2 | 1 | 0 | 0 | 5
  High Grade B Cell Lymphoma | 0 | 0 | 0 | 2 | 1 | 3
  Primary Mediastinal Large B Cell Lymphoma | 0 | 0 | 0 | 0 | 1 | 1
  Nodal marginal zone lymphoma | 1 | 0 | 0 | 0 | 0 | 1
  Follicular lymphoma | 0 | 1 | 2 | 2 | 5 | 10
  Missing | 0 | 0 | 0 | 0 | 1 | 1
International Prognostic Index [Count of Participants; unit: Participants]
  Low risk | 1 | 1 | 1 | 2 | 3 | 8
  Low-intermediate risk | 1 | 2 | 1 | 3 | 9 | 16
  High-intermediate risk | 2 | 0 | 3 | 6 | 2 | 13
  High risk | 0 | 0 | 0 | 5 | 5 | 10
  Not done/Unknown | 0 | 0 | 3 | 1 | 1 | 5
Molecular Subtype [Count of Participants; unit: Participants]
  No High Risk Molecular Features | 2 | 2 | 2 | 6 | 3 | 15
  ouble Hit (myc/bcl2 or myc/bcl6 rearrangement) | 0 | 0 | 4 | 4 | 6 | 14
  Triple Hit (myc/bcl2/bcl6 rearrangement) | 0 | 0 | 0 | 4 | 1 | 5
  Double Expressor (myc and bcl2 overexpression) | 0 | 1 | 1 | 3 | 3 | 8
  Not done/Unknown | 2 | 0 | 1 | 0 | 7 | 10
Sum of Product of Perpendicular Diameters [Median (Full Range); unit: cm] — Last non-missing value prior to pre-conditioning. Population: Data were missing for 3 patients
  cm
    number analyzed (Participants) | 3 | 3 | 7 | 16 | 20 | 49
    (all) | 17.91 [7.0 to 18.7] | 19.31 [17.4 to 48.2] | 28.55 [2.6 to 260.8] | 21.54 [2.1 to 130.3] | 13.19 [2.9 to 163.1] | 18.69 [2.1 to 260.8]
Lactate Dehydrogenase [Median (Full Range); unit: U/L] — Last non-missing value prior to pre-conditioning.
  U/L | 331.50 [228.0 to 664.0] | 403.00 [220.0 to 442.0] | 262.00 [162.0 to 498.0] | 231.00 [132.0 to 1348.0] | 235.00 [156.0 to 1340.0] | 243.50 [132.0 to 1348.0]
Lines of therapy [Median (Full Range); unit: Lines of therapy] | 2.5 [2 to 4] | 3.0 [2 to 4] | 3.0 [2 to 10] | 3.0 [1 to 5] | 3.0 [1 to 6] | 3.0 [1 to 10]
Prior stem cell transplantation [Count of Participants; unit: Participants] | 0 | 1 | 2 | 3 | 10 | 16

OUTCOME MEASURES:

1. Primary Outcome: Phase I Escalation - Safety (Number of Participants With Grade 3-5 Toxicities) and Identification of Recommended Phase II Dose and Schedule (RP2D).
Description: Number of patients with Grade 3-5 toxicities during escalation part of Phase I (Cohorts: 50x10^6 CD19/22 CAR+ T Cells; 50x10^6 CD19/22 CAR+ T Cells+Pembrolizumab [Pem] Day 14; 150-450x10^6 CD19/22 CAR+ T Cells+Pem Day 14; 150-450x10^6 CD19/22 CAR+ T Cells+Pem Day -1 in Inpatient Setting)
  Dose-limiting toxicity defined as:
  * New non-hematological AE Grade >=3 using NCI CTCAE (5.0), probably/definitely related to AUTO3, occurring in DLT evaluation period, which did not resolve to Grade 2 or better in 14 days, despite supportive measures.
  * Grade 4 CRS, neurotoxicity (NT), or cerebral edema, or Grade 3 NT that lasted >72 hrs
  * Grade >3 Disseminated Intravascular Coagulation
  * Grade >2 Infusion Reaction with AUTO3
  * Grade 4 or 5 event not managed with conventional supportive measures or necessitating dose reduction or modification to trial therapy
  * Any event that in opinion of Investigator and/or medical monitor put patient at undue risk could also have been considered DLT
Time Frame: Within 75 days of AUTO3 infusion
Population: Patients who received at least 1 (complete or partial) dose of AUTO3 (infused set)
Measure: Number; unit: participants
Groups:
- 50 x 10^6 CD19/CD22 CAR+ T Cells: Patients in this cohort received actual doses of 50 to 150 x 10^6 CD19/CD22 CAR+ T cells
Arm/Group | 50 x 10^6 CD19/CD22 CAR+ T Cells | 50 x 10^6 CD19/CD22 CAR+ T Cells + Pembrolizumab at Day 14 | 150 to 450 x 10^6 CD19/CD22 CAR+ T Cells + Pembrolizumab at Day 14 | 150 to 450 x 10^6 CD19/CD22 CAR+ T Cells + Pembrolizumab at Day -1 in an Inpatient Setting | 150 to 450 x 10^6 CD19/CD22 CAR+ T Cells + Pembrolizumab at Day -1 in an Outpatient Setting
Number analyzed (Participants) | 4 | 3 | 8 | 17 | 0
participants
  Patients with Grade 3-5 toxicity | 4 | 3 | 7 | 13 |
  Patients with dose-limiting toxicity | 0 | 0 | 0 | 0 |

2. Primary Outcome: Phase I Expansion - Safety (Incidence of Grade 3-5 Toxicities) in the Outpatient / Ambulatory Care Setting
Description: The incidence of Grade 3-5 toxicities during the expansion part of Phase I (Dose cohort: 150 to 450 x 10^6 CD19/CD22 CAR-positive T Cells + Pembrolizumab at Day -1 in an Outpatient Setting)
Time Frame: Within 75 days of AUTO3 infusion
Population: Patients who received at least 1 (complete or partial) dose of AUTO3 (infused set)
Measure: Count of Participants; unit: Participants
Groups:
- 50 x 10^6 CD19/CD22 CAR-positive T Cells: Patients in this cohort received actual doses of 50 to 150 x 10^6 CD19/CD22 CAR-positive T cells
Arm/Group | 50 x 10^6 CD19/CD22 CAR-positive T Cells | 50 x 10^6 CD19/CD22 CAR-positive T Cells + Pembrolizumab at Day 14 | 150 to 450 x 10^6 CD19/CD22 CAR-positive T Cells + Pembrolizumab at Day 14 | 150 to 450 x 10^6 CD19/CD22 CAR-positive T Cells + Pembrolizumab at Day -1 in an Inpatient Setting | 150 to 450 x 10^6 CD19/CD22 CAR-positive T Cells + Pembrolizumab at Day -1 in an Outpatient Setting
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 20
Participants | 0 | 0 | 0 | 0 | 13

3. Primary Outcome: Phase II - Overall Response Rate as Per Lugano Criteria
Description: This was not analysed due to study termination prior to initiation of Phase II. End of study notification submitted to Medicines and Healthcare products Regulatory Agency (MHRA) (reference 46113/0003/001-0016) - The Last patient last visit was 19 October 2023 (at end of Phase 1) and the study is considered completed (End of study). As per protocol v10.0, end of study is defined as 36 months after the last patient has received AUTO3 infusion or earlier in the event of death or consent withdrawal. Fifty-two patients received AUTO3 in the Phase I part of the study. After reviewing the data and taking into consideration the available treatment landscape in r/r DLBCL, Autolus didn't progress AUTO3-DB1 into the Phase II part of the study. Autolus notified MHRA on 08 November 2021 about enrolment to Phase II of the study (Autolus has decided not to progress AUTO3-DB1 into the Phase II part of the study), and MHRA acknowledged it on 09 November 2021.
Time Frame: Up to 2 years
Population: This was not evaluated because no dose-limiting toxicities occurred in the Phase 1 part of the study to identify the recommended dose
Groups:
- Recommended Phase 2 Dose: This was not evaluated because no dose-limiting toxicities occurred in the Phase 1 part of the study to identify the recommended dose. The study was terminated at the end of Phase 1.
Arm/Group | Recommended Phase 2 Dose
Number analyzed (Participants) | 0

4. Secondary Outcome: Feasibility of Generating AUTO3: Number of Patients' Cells Successfully Manufactured as a Proportion of the Number of Patients Undergoing Leukapheresis.
Description: Feasibility of product generation was examined by assessing the number of AUTO3 successfully manufactured as a fraction of the number of patients undergoing leukapheresis (all patients enrolled).
Time Frame: Up to 8 weeks post leukapheresis.
Population: Patients who underwent leukapheresis. This outcome is measured before patients received infusion with AUTO3. Therefore, no split by dose cohort can be provided.
Measure: Count of Participants; unit: Participants
Groups:
- AUTO3: Patient with relapsed or refractory DLBCL
  AUTO3: Following preconditioning with chemotherapy (cyclophosphamide and fludarabine) patients will be treated with doses from 50 x 10⁶ to 900 x 10⁶ CD19/ CD22 Chimeric Antigen Receptor (CAR) positive T cells followed by limited duration of anti-programmed cell death protein (PD)-1 antibody (pembrolizumab).
Arm/Group | AUTO3
Number analyzed (Participants) | 62
Participants | 52

5. Secondary Outcome: Determine the Complete Response Rate Following Treatment With AUTO3, as Per Lugano Criteria.
Description: Participants achieving objective response per Lugano criteria based on independent central radiology review.
  The Lugano classification of response by 18F-2-fluoro-2-deoxy-D-glucose fluorodeoxyglucose (FDG) PET-CT:
  1. no uptake or no residual uptake (when used interim)
  2. slight uptake, but below blood pool (mediastinum)
  3. uptake above mediastinal, but below or equal to uptake in the liver
  4. uptake slightly to moderately higher than liver
  5. markedly increased uptake or any new lesion (on response evaluation) Non-progressive disease
     * complete metabolic response - score of 1, 2 or 3 in nodal or extranodal sites with or without a residual mass
     * partial metabolic response - score of 4 or 5 with reduced uptake compared with baseline and residual mass(es) of any size
     * stable disease or no metabolic response - score of 4 or 5 with no obvious change in FDG uptake Progressive disease score 4 or 5 in any lesion with an increase in intensity of FDG uptake from baseline (and/or
Time Frame: Up to 2 years
Population: All participants who received at least one dose of AUTO3. Five patients had no positive disease by FDG PET scan prior to pre-conditioning (1 in the 50 x 10^6 group, 1 in the 150-450 x 10^6 inpatient group, and 3 in the 15-450 x 10^6 outpatient group). Hence, they were not evaluable for best overall response.
Measure: Count of Participants; unit: Participants
Arm/Group | 50 x 10^6 CD19/CD22 CAR-positive T Cells | 50 x 10^6 CD19/CD22 CAR-positive T Cells + Pembrolizumab at Day 14 | 150 to 450 x 10^6 CD19/CD22 CAR-positive T Cells + Pembrolizumab at Day 14 | 150 to 450 x 10^6 CD19/CD22 CAR-positive T Cells + Pembrolizumab at Day -1 in an Inpatient Setting | 150 to 450 x 10^6 CD19/CD22 CAR-positive T Cells + Pembrolizumab at Day -1 in an Outpatient Setting
Number analyzed (Participants) | 4 | 2 | 8 | 16 | 17
Participants | 1 | 1 | 4 | 8 | 8

6. Secondary Outcome: Duration of Response (DOR).
Description: Duration of response was defined as the time from the first observed complete response or partial response [from the first post-baseline response assessment] until the date of first progressive disease or death due to underlying cancer (primary reason for death=progressive disease), whichever occurred first.
  Only responders (patients with complete response [CR] or partial response [PR]) were included in the analysis of duration of response.
  Response defined by Lugano classification (see Outcome Measure 5). Patients with death not due to underling cancer (primary reason for death=adverse event [AE] or Other or Unknown) or who received new anti-cancer therapy other than SCT or discontinued from the study for other reason than progressive disease (PD) or who were lost to follow-up or reached the time point of analysis without a known record of progression or death had the duration of response censored at the date of last adequate disease assessment for response.
Time Frame: Up to 2 years
Population: Patients who received at least 1 (complete or partial) dose of AUTO3 (infused set). Patients with death not due to underling cancer or who received new anti-cancer therapy other than SCT or discontinued from the study for other reason than progressive disease (PD) or who were lost to follow-up or reached the time point of analysis without a known record of progression or death had the duration of response censored at the date of last adequate disease assessment for response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 50 x 10^6 CD19/CD22 CAR-positive T Cells | 50 x 10^6 CD19/CD22 CAR-positive T Cells + Pembrolizumab at Day 14 | 150 to 450 x 10^6 CD19/CD22 CAR-positive T Cells + Pembrolizumab at Day 14 | 150 to 450 x 10^6 CD19/CD22 CAR-positive T Cells + Pembrolizumab at Day -1 in an Inpatient Setting | 150 to 450 x 10^6 CD19/CD22 CAR-positive T Cells + Pembrolizumab at Day -1 in an Outpatient Setting
Number analyzed (Participants) | 2 | 2 | 5 | 11 | 15
months | 6.31 [1.97 to NA] — Upper limit of the confidence interval was not reached due to insufficient number of events. | NA [NA to NA] — Median estimates and corresponding 95% confidence intervals are not available due to limited number of events and/or insufficient follow-up, which precludes reliable estimation of survival probabilities or confidence intervals using the Kaplan-Meier method. | NA [NA to NA] — Median estimates and corresponding 95% confidence intervals are not available due to limited number of events and/or insufficient follow-up, which precludes reliable estimation of survival probabilities or confidence intervals using the Kaplan-Meier method. | 4.96 [1.91 to NA] — Upper limit of the confidence interval was not reached due to insufficient number of events. | NA [NA to NA] — Median estimates and corresponding 95% confidence intervals are not available due to limited number of events and/or insufficient follow-up, which precludes reliable estimation of survival probabilities or confidence intervals using the Kaplan-Meier method.

7. Secondary Outcome: Progression-free Survival (PFS).
Description: The progression-free survival was defined as the time from first AUTO3 treatment until the first progression of disease or death from any cause, whichever occurred first.
  Patients who reached the time point of analysis without a known record of progression had the PFS censored at the date of last adequate disease assessment.
  Patients who received a new stem cell transplantation (SCT) were censored at the start date of this new SCT.
  Patients who received a new anti-cancer therapy or discontinued from the study for other reason than disease progression and who were lost to follow-up were censored at the date of last adequate disease assessment.
  Response defined by Lugano classification (see Outcome Measure 5).
Time Frame: Up to 2 years
Population: Patients who received at least 1 (complete or partial) dose of AUTO3 (infused set) and were not censored.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 50 x 10^6 CD19/CD22 CAR-positive T Cells | 50 x 10^6 CD19/CD22 CAR-positive T Cells + Pembrolizumab at Day 14 | 150 to 450 x 10^6 CD19/CD22 CAR-positive T Cells + Pembrolizumab at Day 14 | 150 to 450 x 10^6 CD19/CD22 CAR-positive T Cells + Pembrolizumab at Day -1 in an Inpatient Setting | 150 to 450 x 10^6 CD19/CD22 CAR-positive T Cells + Pembrolizumab at Day -1 in an Outpatient Setting
Number analyzed (Participants) | 4 | 3 | 8 | 17 | 20
months | 2.14 [0.76 to NA] — Upper limit of the confidence interval was not reached due to insufficient number of events. | 2.43 [2.40 to NA] — Upper limit of the confidence interval was not reached due to insufficient number of events. | 5.67 [0.95 to NA] — Upper limit of the confidence interval was not reached due to insufficient number of events. | 3.22 [1.87 to NA] — Upper limit of the confidence interval was not reached due to insufficient number of events. | 3.22 [1.94 to 5.88]

8. Secondary Outcome: Overall Survival (OS).
Description: Overall survival (OS) was defined as the time from the date of first AUTO3 treatment up to the date of death, regardless of cause of death.
  Patients alive at the time of the analysis had the OS censored at the date of last assessment when the patient was known alive.
Time Frame: Up to 2 years
Population: Patients who received at least 1 (complete or partial) dose of AUTO3 (infused set) and were not censored.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 50 x 10^6 CD19/CD22 CAR-positive T Cells | 50 x 10^6 CD19/CD22 CAR-positive T Cells + Pembrolizumab at Day 14 | 150 to 450 x 10^6 CD19/CD22 CAR-positive T Cells + Pembrolizumab at Day 14 | 150 to 450 x 10^6 CD19/CD22 CAR-positive T Cells + Pembrolizumab at Day -1 in an Inpatient Setting | 150 to 450 x 10^6 CD19/CD22 CAR-positive T Cells + Pembrolizumab at Day -1 in an Outpatient Setting
Number analyzed (Participants) | 4 | 3 | 8 | 17 | 20
months | 10.04 [0.95 to NA] — Upper limit of the confidence interval was not reached due to insufficient number of events. | 6.67 [4.93 to NA] — Upper limit of the confidence interval was not reached due to insufficient number of events. | 5.67 [1.77 to NA] — Upper limit of the confidence interval was not reached due to insufficient number of events. | 9.17 [3.32 to NA] — Upper limit of the confidence interval was not reached due to insufficient number of events. | NA [NA to NA] — Median estimates and corresponding 95% confidence intervals are not available due to limited number of events and/or insufficient follow-up, which precludes reliable estimation of survival probabilities or confidence intervals using the Kaplan-Meier method.

9. Other Pre Specified Outcome: To Determine the Expansion and Persistence of AUTO3 Following Adoptive Transfer in Different Lymphoma Subtypes (Maximum Concentration)
Description: Analysis of cells in peripheral blood by polymerase chain reaction and/or flow cytometry at a range of time points in the peripheral blood.
Time Frame: Up to 2 years
Population: Patients who received at least 1 (complete or partial) dose of AUTO3 (infused set).
Measure: Geometric Mean (Full Range); unit: copies/microgram DNA
Arm/Group | 50 x 10^6 CD19/CD22 CAR-positive T Cells | 50 x 10^6 CD19/CD22 CAR-positive T Cells + Pembrolizumab at Day 14 | 150 to 450 x 10^6 CD19/CD22 CAR-positive T Cells + Pembrolizumab at Day 14 | 150 to 450 x 10^6 CD19/CD22 CAR-positive T Cells + Pembrolizumab at Day -1 in an Inpatient Setting | 150 to 450 x 10^6 CD19/CD22 CAR-positive T Cells + Pembrolizumab at Day -1 in an Outpatient Setting
Number analyzed (Participants) | 4 | 3 | 7 | 17 | 20
copies/microgram DNA | 7979.7 [155 to 213000] | 13157.4 [3900 to 47100] | 5726.1 [1420 to 11600] | 4121.4 [174 to 416000] | 3195.6 [241 to 131000]

10. Other Pre Specified Outcome: To Determine the Expansion and Persistence of AUTO3 Following Adoptive Transfer in Different Lymphoma Subtypes (Area Under the Curve From Day 0 to Day 28)
Description: as for outcome 9
Time Frame: Up to 2 years
Population: Patients who received at least 1 (complete or partial) dose of AUTO3 (infused set).
Measure: Geometric Mean (Full Range); unit: day*copies/microgram DNA
Arm/Group | 50 x 10^6 CD19/CD22 CAR-positive T Cells | 50 x 10^6 CD19/CD22 CAR-positive T Cells + Pembrolizumab at Day 14 | 150 to 450 x 10^6 CD19/CD22 CAR-positive T Cells + Pembrolizumab at Day 14 | 150 to 450 x 10^6 CD19/CD22 CAR-positive T Cells + Pembrolizumab at Day -1 in an Inpatient Setting | 150 to 450 x 10^6 CD19/CD22 CAR-positive T Cells + Pembrolizumab at Day -1 in an Outpatient Setting
Number analyzed (Participants) | 4 | 3 | 7 | 17 | 20
day*copies/microgram DNA | 41511.0 [912 to 2370000] | 109945.2 [35600 to 478000] | 38397.9 [3510 to 135000] | 37722.7 [948 to 571000] | 32152.1 [1060 to 1930000]

11. Other Pre Specified Outcome: To Determine the Expansion and Persistence of AUTO3 Following Adoptive Transfer in Different Lymphoma Subtypes (Time to Maximum Concentration)
Description: as for outcome 9
Time Frame: Up to 2 years
Population: Patients who received at least 1 (complete or partial) dose of AUTO3 (infused set).
Measure: Median (Full Range); unit: Days
Arm/Group | 50 x 10^6 CD19/CD22 CAR-positive T Cells | 50 x 10^6 CD19/CD22 CAR-positive T Cells + Pembrolizumab at Day 14 | 150 to 450 x 10^6 CD19/CD22 CAR-positive T Cells + Pembrolizumab at Day 14 | 150 to 450 x 10^6 CD19/CD22 CAR-positive T Cells + Pembrolizumab at Day -1 in an Inpatient Setting | 150 to 450 x 10^6 CD19/CD22 CAR-positive T Cells + Pembrolizumab at Day -1 in an Outpatient Setting
Number analyzed (Participants) | 4 | 3 | 7 | 17 | 20
Days | 16.4 [12 to 22] | 13.9 [11 to 14] | 9.7 [9 to 35] | 10.0 [7 to 28] | 13.1 [7 to 58]

ADVERSE EVENTS:
Time Frame: From AUTO3 infusion (Day -7) until end of study/patient withdrawal OR, when patient initiated a new treatment for their disease (approximately 3 years and 5 months).
Description: All adverse events (AEs)/serious adverse events (SAEs) were recorded from admission for pre-conditioning chemotherapy (Day -7 relative to AUTO3). Due to the long period between consent and AUTO3 treatment, any AEs/SAEs related to bridging chemotherapy not associated with study procedures did not require reporting as study AEs/SAEs. Any significant events were added to the patient's medical history. All AEs/SAEs related to study procedures (leukapheresis, bone marrow assessments) were reported.
Groups:
- 50 x 10^6 CD19/CD22 CAR+ T Cells: Patients in this cohort received actual doses of 50 to 150 x 10^6 CD19/CD22 CAR-positive T cells
- 50 x 10^6 CD19/CD22 CAR+ T Cells + Pembrolizumab at Day 14: Patients in this cohort received actual dose of 50 x 10^6 CD19/CD22 CAR-positive T cells + pembrolizumab at Day 14
- 150 to 450 x 10^6 CD19/CD22 CAR+ T Cells + Pembrolizumab at Day 14: Patients in this cohort received actual doses of 150 to 495 x 10^6 CD19/CD22 CAR-positive T cells + pembrolizumab at Day 14
- 150 to 450 x 10^6 CD19/CD22 CAR+ T Cells + Pembrolizumab at Day -1 in an Inpatient Setting: Patients in this cohort received actual doses of 125 to 450 x 10^6 CD19/CD22 CAR-positive T cells + pembrolizumab at Day -1 in an inpatient setting
- 150 to 450 x 10^6 CD19/CD22 CAR+ T Cells + Pembrolizumab at Day -1 in an Outpatient Setting: Patients in this cohort received actual doses of 129 to 450 x 10^6 CD19/CD22 CAR-positive T cells + pembrolizumab at Day -1 in an outpatient setting
- Treatment Not Received: Patients enrolled who did not receive study medication
Arm/Group | 50 x 10^6 CD19/CD22 CAR+ T Cells | 50 x 10^6 CD19/CD22 CAR+ T Cells + Pembrolizumab at Day 14 | 150 to 450 x 10^6 CD19/CD22 CAR+ T Cells + Pembrolizumab at Day 14 | 150 to 450 x 10^6 CD19/CD22 CAR+ T Cells + Pembrolizumab at Day -1 in an Inpatient Setting | 150 to 450 x 10^6 CD19/CD22 CAR+ T Cells + Pembrolizumab at Day -1 in an Outpatient Setting | Treatment Not Received
All-Cause Mortality (participants affected / at risk) | 3/4 | 2/3 | 5/8 | 11/17 | 6/20 | 6/10
Serious Adverse Events (participants affected / at risk) | 2/4 | 0/3 | 3/8 | 10/17 | 14/20 | 0/10
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3 | 8/8 | 15/17 | 19/20 | 1/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 50 x 10^6 CD19/CD22 CAR+ T Cells (N=4) | 50 x 10^6 CD19/CD22 CAR+ T Cells + Pembrolizumab at Day 14 (N=3) | 150 to 450 x 10^6 CD19/CD22 CAR+ T Cells + Pembrolizumab at Day 14 (N=8) | 150 to 450 x 10^6 CD19/CD22 CAR+ T Cells + Pembrolizumab at Day -1 in an Inpatient Setting (N=17) | 150 to 450 x 10^6 CD19/CD22 CAR+ T Cells + Pembrolizumab at Day -1 in an Outpatient Setting (N=20) | Treatment Not Received (N=10)
Abdominal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 1 | 0 | 1 | 1 | 5 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Enterobacter infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Enterococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Facial paresis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 2 | 3 | 0
Gallbladder abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Immune effector cell-associated neurotoxicity syndrome (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nystagmus (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 2 | 0 | 0 | 2 | 3 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Actinomycotic pulmonary infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Colitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0
Device related infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 0 | 0 | 1 | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Nervous system disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Parkinson's disease (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 50 x 10^6 CD19/CD22 CAR+ T Cells (N=4) | 50 x 10^6 CD19/CD22 CAR+ T Cells + Pembrolizumab at Day 14 (N=3) | 150 to 450 x 10^6 CD19/CD22 CAR+ T Cells + Pembrolizumab at Day 14 (N=8) | 150 to 450 x 10^6 CD19/CD22 CAR+ T Cells + Pembrolizumab at Day -1 in an Inpatient Setting (N=17) | 150 to 450 x 10^6 CD19/CD22 CAR+ T Cells + Pembrolizumab at Day -1 in an Outpatient Setting (N=20) | Treatment Not Received (N=10)
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 1 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 6 | 9 | 8 | 0
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Anal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Application site vesicles (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Autonomic nervous system imbalance (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 3 | 0
Blood fibrinogen decreased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Blood lactic acid increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Blood phosphorus decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Blood potassium decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Blood uric acid decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Burn oral cavity (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Catheter site infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Catheter site inflammation (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 1 | 4 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 2 | 2 | 5 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 2 | 0 | 3 | 4 | 5 | 0
Cytomegalovirus test positive (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis psoriasiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Device related thrombosis (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 2 | 2 | 4 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 5 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dysmetria (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 3 | 1 | 0
Ear discomfort (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Enterococcal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Epigastric discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 3 | 0
Fatigue (General disorders) | 1 | 1 | 4 | 2 | 8 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 2 | 1 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Gallbladder enlargement (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hallucination, visual (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 0 | 5 | 2 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hyperferritinaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0
Hypogammaglobulinaemia (Immune system disorders) | 0 | 0 | 1 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 2 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 1 | 1 | 1 | 2 | 0
Hypotension (Vascular disorders) | 1 | 0 | 4 | 0 | 2 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 3 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Lymph node pain (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 3 | 0
Malaise (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 2 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 1 | 2 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 4 | 9 | 5 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 4 | 3 | 3 | 3 | 2 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 1 | 0 | 0
Ocular icterus (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 1 | 4 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 2 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Osteosclerosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 2 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0
Pancreatic mass (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0
Parvovirus infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Physical deconditioning (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Platelet count decreased (Investigations) | 4 | 3 | 3 | 2 | 4 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 2 | 4 | 1 | 5 | 0
Radiation skin injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1 | 0 | 0
Rash maculo-papular (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 2 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Rash pustular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Respiratory alkalosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Serum ferritin increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Staphylococcal abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Staphylococcal infection (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
Superinfection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 1 | 1 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Taste disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Tension headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Terminal ileitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 7 | 3 | 0
Thrombosis in device (Product Issues) | 0 | 0 | 0 | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vaginal fistula (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vascular device occlusion (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 2 | 0 | 2 | 0
Weight decreased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0
Weight increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 2 | 0 | 4 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hepatitis B reactivation (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Myocarditis (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Parkinson's disease (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pharyngitis bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Only results of Phase I of the study are presented due to study termination prior to initiation of Phase II.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-05-06): https://cdn.clinicaltrials.gov/large-docs/17/NCT03287817/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-21): https://cdn.clinicaltrials.gov/large-docs/17/NCT03287817/SAP_001.pdf